CLINICAL TRIAL: NCT07244107
Title: Comparative Effects of FIFA 11+ and RAMP Protocols on Agility and Sprint Performance Outcomes in Young Soccer Players
Brief Title: Agility and Sprint Performance in Youth Soccer: A Comparison of FIFA 11+ and RAMP Protocols
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/ADILMUNIR
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Children, Adult
Keywords: Youth soccer; Warm-up protocols; FIFA 11+; RAMP; Agility; Sprint

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial (RCT) designed to compare the effectiveness of two different warm-up routines on the physical performance of young soccer players. The study will involve 34 male participants between the ages of 8 and 15. These participants will be randomly divided into two groups. One group will follow the FIFA 11+ protocol, a warm-up designed for injury prevention and neuromuscular control, which consists of specific running, strength, and balance exercises. The other group will use the RAMP protocol, which systematically prepares athletes for high-intensity activity through four phases: Raise, Activate, Mobilize, and Potentiate. The trial will last for six weeks, with performance in agility and sprinting measured before and after the intervention to determine which protocol yields greater improvements.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ Protocol Group (Active Comparator): Participants in this group will perform the FIFA 11+ warm-up protocol at the beginning of each training session for six weeks. This comprehensive, 20-minute program consists of 15 exercises, 3 days a week. Participants with receive total 18 sessions.
  Interventions: Other: FIFA 11+ Warm-Up Program
- RAMP Protocol Group (Active Comparator): Participants in this group will perform the RAMP warm-up protocol at the beginning of each training session for six weeks. This protocol is a systematic, four-phase approach designed to progressively prepare athletes for high-intensity activity, 20 minutes session, 3 days a week. Participants with receive total 18 sessions.
  Interventions: Other: RAMP Warm-Up Program

INTERVENTIONS:
Other: FIFA 11+ Warm-Up Program — The intervention for the first group is the FIFA 11+ warm-up protocol, a standardized 20-minute program developed by FIFA for injury prevention and performance enhancement. It consists of 15 exercises performed in a specific sequence at the start of each training session, divided into three parts: the first part (8 minutes) involves slow-speed running combined with active stretching and partner contacts to practice cutting, deceleration, and proper landing; the second part (10 minutes) focuses on strength, plyometrics, and balance exercises, including core stability, eccentric hamstring strengthening, and proprioceptive training, with three progressive difficulty levels; and the third part (2 minutes) consists of high-intensity running drills with planting and cutting movements to prepare for game-speed activities.
  Arms: FIFA 11+ Protocol Group
Other: RAMP Warm-Up Program — The intervention for the second group is the RAMP (Raise, Activate, Mobilize, Potentiate) protocol, a systematic, four-phase warm-up designed to progressively prepare athletes for high-intensity performance. The first phase, Raise (5 minutes), uses light cardiovascular activities like jogging and skipping to elevate body temperature and heart rate. The second phase, Activate (5 minutes), involves dynamic mobility exercises such as leg swings, lunges, and bodyweight squats to activate key muscle groups. The third phase, Mobilize (5 minutes), focuses on enhancing joint range of motion and movement patterns through dynamic stretches and sport-specific drills. The final phase, Potentiate (5 minutes), includes high-intensity, explosive activities like sprint accelerations, box jumps, and change-of-direction drills to activate the nervous system and optimize neuromuscular readiness for peak performance.
  Arms: RAMP Protocol Group

SUMMARY:
This randomized clinical trial investigates the comparative effects of the FIFA 11+ and RAMP (Raise, Activate, Mobilize, Potentiate) warm-up protocols on the agility and sprint performance of young soccer players. The study involves 34 male players aged 8 to 15, who will be randomly assigned to one of the two warm-up groups for a six-week intervention period. Key performance outcomes-agility, measured by the Illinois Agility Test, and sprint speed, measured by a 30-meter sprint test-will be assessed both before and after the intervention. The research aims to address a gap in sports science by directly comparing these two popular protocols in a youth population, with the goal of providing coaches with clear, evidence-based recommendations for optimizing athlete development and reducing injury risk. Data will be analyzed through SPSS version 27.00.

DETAILED DESCRIPTION:
This randomized clinical trial provides a detailed comparison of the FIFA 11+ and RAMP (Raise, Activate, Mobilize, Potentiate) warm-up protocols to determine their respective impacts on agility and sprint performance in young male soccer players. The study is grounded in the understanding that soccer requires exceptional speed and agility, and that well-structured warm-ups are critical for enhancing performance and preventing injuries, especially during the crucial developmental years of youth athletes. While both FIFA 11+ (a program focused on neuromuscular control and injury prevention) and RAMP (a systematic, four-phase preparation protocol) are widely used, there is a notable lack of research directly comparing their acute effectiveness in a youth soccer context. This study seeks to fill that gap by providing empirical evidence to guide coaches and practitioners in selecting the most effective warm-up strategy.

The study will recruit 34 male soccer players between the ages of 8 and 15, who will be randomly assigned to either the FIFA 11+ or the RAMP intervention group for a six-week period. Performance will be measured using standardized, valid, and reliable tests: the Illinois Agility Test (IAT) to assess agility and a 30-meter sprint test to measure speed. These assessments will be conducted at baseline before the intervention begins and again immediately following the six-week training period. The collected data will be analyzed to compare within-group improvements and between-group differences, with statistical adjustments for baseline values to ensure a robust comparison. The findings are expected to offer practical, evidence-based recommendations for optimizing warm-up routines to specifically enhance agility and sprint capabilities in young soccer players, thereby supporting superior athletic development. Data will be analyzed through SPSS version 27.00.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 8-15 years.
* Minimum one year of organized soccer experience.
* Currently training at least three times per week.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Cardiovascular, neurological, or musculoskeletal disorders.
* Musculoskeletal injury in the past six months.
* Participation in other structured injury prevention or strength programs.
* Inability to complete baseline testing.

Ages: 8 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — This study is limited to male participants only. The focus on a single gender is intended to reduce potential confounding variables related to sex-based differences in physiological development, neuromuscular control, and response to training during adolescence. By restricting the study population to males, the research aims to achieve a more homogenous sample, thereby increasing the internal validity of the comparison between the FIFA 11+ and RAMP warm-up protocols.
Enrollment: 34 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Illinois Agility Test (IAT) | [Time Frame: Baseline, 1st week and 6th week]
  The Illinois Agility Test is a field-based assessment designed to measure an athlete's ability to accelerate, decelerate, and change direction rapidly. The test involves sprinting and weaving through a set course marked by cones. The total time to complete the course is recorded using a stopwatch. The IAT is a highly valid and reliable tool for assessing agility. Recent studies report high content validity (Aiken's V = 0.93) and strong reliability (r = 0.81), confirming its effectiveness for evaluating agility in athletes. Additional research has shown the IAT to have excellent interrater reliability and moderate to good test-retest reliability, making it suitable for both research and applied sports settings.
Stopwatch for Sprint Speed | [Time Frame: Baseline, 1st week and 6th week]
  A standard handheld stopwatch is used to measure sprint speed over set distance 30m. The assessor starts and stops the watch as the participant crosses the start and finish lines. The best time from two trials is recorded for analysis. Manual timing with a stopwatch is a practical and cost-effective method for field-based sprint assessment. Research shows that hand-held stopwatches have strong concurrent validity compared to electronic timing systems (R² = 0.981-0.994) and excellent inter-rater reliability (ICC = 0.980-0.994) when used by experienced raters. The typical measurement error is small (about 1.6-2.5%), making this method acceptable for sports performance testing.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Munir, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Model Town Football Club, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panchal R, Rizvi MR, Sharma A, Ahmad F, Hasan S, Shaik AR, Seyam MK, Uddin S, Ahamed WM, Iqbal A, Alghadir AH. Comparing the effectiveness of the FIFA 11+ warm-up and conventional warm-up in enhancing cyclist performance and mitigating injury risk. Sci Rep. 2025 Mar 19;15(1):9430. doi: 10.1038/s41598-025-91005-z. PMID 40108222